CLINICAL TRIAL: NCT02272894
Title: Randomized Controlled Trial to Evaluate Mesenteric Vein (14V) Lymphadenectomy for Gastric Cancer
Brief Title: A Trial to Evaluate the Superior Mesenteric Vein (14V) Lymphadenectomy for Distal Advanced Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Shanxi Province Cancer Hospital (Other); Peking University Cancer Hospital & Institute (Other); Qingdao University (Other); Fudan University (Other); Sun Yat-sen University (Other); Harbin Medical University (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); The First Affiliated Hospital of Dalian Medical University (Other); Qinghai University (Other); Second Hospital of Jilin University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Wulumuqi General Hospital of Lanzhou Military Command (Other); Shandong Provincial Hospital (Other Government); Nanjing PLA General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: E201419A
Record Dates: First submitted 2014-09-15; First posted 2014-10-23 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2014-07

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; D2 Lymphadenectomy; Superior Mesenteric Vein Lymph Node
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group A: D2 Radical Gastrectomy Adding Dissection of the Superior Mesenteric Vein Lymph Node
  Interventions: Procedure: Dissection of the Superior Mesenteric Vein Lymph Node
- Group B: D2 Radical Gastrectomy

INTERVENTIONS:
Procedure: Dissection of the Superior Mesenteric Vein Lymph Node — 14v lymph node dissection
  Groups: Group A

SUMMARY:
This trial is going to evaluate the advantage of D2 radical gastrectomy plus 14v lymph node dissection in 3-year survival rates of advanced gastric cancers.

DETAILED DESCRIPTION:
Radical surgery is still the only possible way to cure gastric cancer. In Japan, South Korea and other countries, due to the popularity of screening and Improved surgical procedures, there has been great improvement in overall survival. Standard D2 Gastrectomy has been the standard operation for advanced gastric cancer. However, there is no unanimous consensus whether Standard D2 Gastrectomy plus 14v lymph node dissection is needed.Till now, it is difficult to stage the 14V lymph node as regional lymph nodes metastasis or distant metastasis. And it is urgent to explore the necessity of 14v lymph node dissection in advanced gastric cancer.So a prospective randomized controlled study will to carry out to evaluate the effects of D2 radical gastrectomy plus 14v lymph node dissection compared with D2 radical gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Curative D2 or D2+ operation had been performed;
* Physical condition and organ function allows to tolerable abdominal surgery;
* Willing and able to comply with the program during the study period;
* Aged 18 to 70 years, preoperative gastric cancer patients with pathologically confirmed;
* With more than a 6-month life expectancy;
* No other serious concomitant diseases;
* No adjuvant chemotherapy before recurrence;
* Karnofsky performance status scale ≥ 60;
* All patients accept 6 cycles XELOX chemotherapy regimen

Exclusion Criteria:

* Pregnancy or breast feeding;
* Women of childbearing age do not take contraceptive measures;
* Organ transplantation patients need immunosuppressive therapy;
* Five years after the trial begin,other malignant tumor occur;
* While using other experimental drug or other clinical trials are being;
* Can not take oral medications;
* Mentally disordered;
* Severe recurrent infections were not controlled or with other serious concomitant diseases;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Distal Advanced Gastric Cancer
Sampling Method: Probability Sample
Enrollment: 510 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 years
  Overall survival (OS) was defined as the length of time from the date of randomization to the date of death of various reasons.

SECONDARY OUTCOMES:
disease free survival | 3 years
  Disease free survival (DFS) was defined as the length of time from the date of randomization to the date of first documentation of relapse of gastric cancer or any other type of cancer or death.

CONTACTS AND LOCATIONS:
Overall Officials: Han Liang, Master, Principal Investigator — Tianjin Medical University Cancer Hospital
Locations (1):
- Department of Gastrointestinal Medical Oncology, Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Yang QC, Zhou HK, Yue C, Wang WD, Gao RQ, Mo ZC, Ji PP, Wei JP, Yang XS, Yu PF, Li XH, Ji G. [The correlation between No. 6 and No. 14v lymph node metastasis and the value of dissecting these lymph nodes in radical gastrectomy]. Zhonghua Wei Chang Wai Ke Za Zhi. 2023 Jan 25;26(1):38-43. doi: 10.3760/cma.j.cn441530-20221123-00491. Chinese. PMID 36649998